CLINICAL TRIAL: NCT01549912
Title: Results of Rotator Cuff Repair Following Acute Shoulder Dislocation
Brief Title: Results of Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Tashjian, M.D., University of Utah
Other Study IDs: 54314
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Shoulder Dislocation
Keywords: Rotator Cuff Tears; Dislocation; Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation; Rotator Cuff Injuries; Joint Dislocations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rotator cuff tear

SUMMARY:
The primary objective of this research is to examine the result of rotator cuff repairs following acute shoulder dislocations and to investigate whether timing of surgery following acute shoulder dislocations affects patients perception of pain, function, and strength following surgery.

DETAILED DESCRIPTION:
There is a higher risk of rotator cuff tears following dislocation when the individual is greater than 40 years old. Rotator cuff tears after dislocation of the shoulder are more of a challenge to repair particularly if there is a delay in diagnosis. Clinical experience would suggest that rotator cuff repair within the first month of injury allows for better results in acute rotator cuff tears without shoulder dislocation. There are no reported results for rotator cuff repairs following shoulder dislocation and timing of repair. If we find that early repair provides better results this will be important for Primary Care Providers and Emergency Department physicians to refer these patients early for evaluation and subsequently earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 35 years or older with acute rotator cuff tear following documented shoulder dislocation requiring reduction, subjects sustained acute rotator cuff tear following shoulder dislocation that was treated surgically with open and/or arthroscopic technique between January 1, 2001 and June 1, 2011, surgical intervention within 6 months of dislocation, minimum follow up time of one year from surgery.

Exclusion Criteria:

* rotator cuff tears without shoulder dislocation, known previous rotator cuff disease, history of other trauma to the shoulder, inability to provide informed consent, other suspect pathology (ie: tumor, infection).

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include patients age 35 years and older who have sustained an acute rotator cuff tear following shoulder dislocation who underwent a rotator cuff repair either by open or arthroscopic techniques between January 1, 2001 and June 1, 2011.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Levels of pain, range of motion and strength | 1 year
  Patient are asked to complete ASES, SST, SF-12 questionaires. Clinical evaluation of bilateral range of motion and strength measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Z Tashjian, MD, Principal Investigator — University of Utah Orthopaedic
Locations (1):
- University of Utah, Salt Lake City, Utah, United States